CLINICAL TRIAL: NCT00564096
Title: A Prospective Multicenter Double Blind Randomized Controlled Trial to Explore the Tolerability, Safety and Efficacy of the H1-Coil Deep Transcranial Magnetic Stimulation (TMS) in Subjects With Schizophrenia Experiencing Auditory Hallucinations
Brief Title: Transcranial Magnetic Stimulation (TMS) in Schizophrenia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Dr. Oded Rosenberg, Beer Yaakov
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TMS-218CTIL; HT4413
Record Dates: First submitted 2007-11-25; First posted 2007-11-27 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2009-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real TMS (Active Comparator): 10 patients will be given 20 minutes stimulation with real deep H1-Coil TMS to the Left Temporo-parietal Cortex in frequency of 1 Hz with 120% motor threshold during 20 consecutive working days.
  Interventions: Device: DEEP TMS H1 coil
- Sham & real TMS (Placebo Comparator): 10 patients will be given 20 minutes stimulation with sham deep H1-Coil TMS to the Left Temporo-parietal Cortex in frequency of 1 Hz with 120% motor threshold during 10 consecutive working days, and thereafter 20 sessions of real TMS with the same parameters (=Left Tempor-oparietal Cortex in frequency of 1 Hz with 120% motor threshold).
  Interventions: Device: Deep H1 coil TMS

INTERVENTIONS:
Device: DEEP TMS H1 coil — A new coil ("H"-coil invented in Weizmann Institute of Science, Neurobiology Department, Rehovot, Israel) capable of stimulating more than twice this depth (Up to 5 cm) was recently developed and hence will be called deep TMS.
  Arms: Real TMS
Device: Deep H1 coil TMS — A new coil ("H"-coil invented in Weizmann Institute of Science, Neurobiology Department, Rehovot, Israel) capable of stimulating more than twice this depth (Up to 5 cm) was recently developed and hence will be called deep TMS.
  Arms: Sham & real TMS

SUMMARY:
Until recently stimulation of nervous tissue deeper than approximately 2 cm from the scalp (will hence be called non-deep TMS) was not possible (3).A new coil ("H"-coil invented in Weizmann Institute of Science, Neurobiology Department, Rehovot, Israel ) capable of stimulating more than twice this depth (Up to 5 cm)was recently developed.Deep TMS is using this h-coil.

Auditory hallucinations are reported by 50% to 70% of patients with schizophrenia and generally consist of spoken speech or "voices." . Patients usually describe the hallucinatory experience as distressing, consistent with evidence that the most common hallucinated utterances are abusive terms,contributing in up to 25% of the cases to a serious suicide attempt.The neuroanatomical basis of auditory hallucinations is thought to involve increasing blood flow of the speech perception areas of the brain, such as the superior temporal cortex of the dominant hemisphere as well as right and left superior temporal cortex.Brain imaging studies of patients with auditory hallucinations have revealed an active area in the right and left superior temporal cortex, Broca's area, and the left temporoparietal cortex. Shergill et al. reported the presence of active areas in the anterior cingulate cortex, right thalamus, left hippocampus, and parahippocampal cortex when subjects were experiencing auditory hallucinations.

Magnetic Stimulation of Left Temporoparietal Cortex suggest that the mechanism of auditory hallucinations involves activation of the left temporoparietal cortex.Reasons to believe that right frontotemporal TMS stimulation cortex can ameliorate auditory hallucinations include evidence that right temporoparietal stimulation achieved significant changes in the frequency of auditory hallucinations,in the patients with auditory hallucinations an increase in blood flow is noted in the right superior temporal gyrus,right temporal lobe activation during auditory hallucination,effect of rTMS can spread to the opposite hemisphere through interhemispheric connections,some evidence that brain circuits involved in the production of auditory hallucinations and symptoms of schizophrenia are widespread and not confined in the left temporoparietal cortex.Deep TMS can reach brain structures as deep as 5 cm whereas non-deep TMS can reach structures less than half that distance. As deep brain structures such as thalamic, limbic and paralimbic regions have been shown to be activated during auditory hallucinations and suspected to play a role in the pathogenesis of auditory hallucinations, their stimulation may attenuate auditory hallucinations. Non-deep TMS can stimulate the cortex but not the neuronal pathways connecting it to deeper brain structures and which stimulation may be additive.

DETAILED DESCRIPTION:
Research of deep TMS treatment in patients with schizophrenia experiencing auditory hallucinations, double blind placebo(sham) controlled study October 14, 2007

Physical background

Modern TMS began in 1985 when Barker and colleagues in Sheffield, UK, developed the first TMS device. However, the original commercially available stimulators were limited in the frequency with which they could produce stimuli by the recharging circuits therefore only allowing for the application of single-pulse TMS. To date, devices capable of stimulating the brain at frequencies up to 100 Hz have opened up new possibilities in magnetic stimulation.

TMS is based on Faraday's principle of electromagnetic induction. A rapidly changing magnetic field (2 T) is generated by passing a very brief (0.2-0.9 milliseconds (ms)) high-current alternating electric pulse through an insulated coil made of wire. When the coil is placed against the scalp the magnetic field passes readily through the skull and induces a weak electrical current in the superficial cortex of the brain lasting exactly as long as the current pulse in the coil. The induced electrical activity can cause cortical neurons to discharge action potentials.Until recently stimulation of nervous tissue deeper than approximately 2 cm from the scalp was not possible.

Neurobiological background

TMS have been proved to modulate a variety of brain substances including increase in the expression of neuropeptide cholecystokinin (CCK) mRNA in rats, increases the firing rate of dopaminergic neurons in the ventral tegmental area and in the substantia nigra,elevation of taurine serine and aspartate in the hypothalamic paraventricular nucleus, release of monoamines in the hippocampus,(which is believed to be highly involved in the pathophysiology of depression), increase in hippocampal serotonin and 5-HIAA content after acute rTMS, a selective increase in 5-HT1A binding sites in the frontal cortex, the cingulated cortex, and the anterior olfactory nucleus in response to a single train of rTMS,as well as down regulation of cortical b-adrenergic receptors.

General clinical background

TMS holds the potential of being able to selectively modulate activity in brain areas involved in pathological processes such as depression, mania, obsessive-compulsive disorder, post-traumatic stress disorder and schizophrenia.

The largest single area of TMS research in psychiatry has been the exploration of possible therapeutic effects of cortical, usually prefrontal, stimulation on symptoms of major depression.

Clinical, neurophysiological and imaging background of auditory hallucinations

Auditory hallucinations are reported by 50% to 70% of patients with schizophrenia and generally consist of spoken speech or "voices." Evidences include review of 16 studies that found an average prevalence of 60% for auditory hallucinations in patients with a diagnosis of schizophrenia. Patients usually describe the hallucinatory experience as distressing, consistent with evidence that the most common hallucinated utterances are abusive terms,contributing in up to 25% of the cases to a serious suicide attempt.

The neuroanatomical basis of auditory hallucinations is thought to involve increasing blood flow of the speech perception areas of the brain, such as the superior temporal cortex of the dominant hemisphere as well as right and left superior temporal cortex.

Brain imaging studies of patients with auditory hallucinations have revealed an active area in the right and left superior temporal cortex, Broca's area, and the left temporoparietal cortex. Shergill et al. reported the presence of active areas in the anterior cingulate cortex, right thalamus, left hippocampus, and parahippocampal cortex when subjects were experiencing auditory hallucinations.

Magnetic Stimulation of Left Temporoparietal Cortex suggest that the mechanism of auditory hallucinations involves activation of the left temporoparietal cortex.

SPET during auditory hallucinations in patients with schizophrenia demonstrated blood flow in the left inferior frontal region (Broca's area) during hallucinations, thus implicating the language-production areas in the experience of auditory hallucinations.Other Positron emission tomography study demonstrated activations in subcortical nuclei (thalamic, striatal), limbic structures (especially hippocampus), and paralimbic regions (parahippocampal and cingulate gyri, as well as orbitofrontal cortex).

TMS based double blind study showed that in auditory hallucinations, the preferentially affected area appears to be located in the primary auditory cortex, rather than the secondary or association areas of the posterior planum temporale.

Positron emission tomography with [18F]-fluorodeoxyglucose in 12 DSM-III schizophrenic patients who experienced auditory hallucinations during glucose uptake compared with the patients who did not experience hallucinations showed that the patients who did experience hallucinations had significantly lower relative metabolism in auditory and Wernicke's regions and a trend toward higher metabolism in the right hemisphere homologue of Broca's region.

Some researchers have suggested that the hallucinated voice might actually be inner speech that is misperceived as stimulation from the outside.

Safety

Generally, the TMS treatment was reported to be well tolerated. No serious adverse effects were reported by any of the patients. There is no evidence that rTMS causes structural brain damage or detrimental cellular alterations. There is however, a low risk of inducing seizures with rTMS and the risk increases with higher stimulation frequencies and intensities. Headache was the main side effect reported,however, the incidence of headaches after approximately 250 treatment sessions, was found to be as high as 8%.

Regarding auditory hallucinations, Safety of TMS when given to Left Temporoparietal Cortex was generally well tolerated with the exception of transient Concentration and memory difficulties lasting 5 to 10 minutes following rTMS ,and that also not more frequently than sham arm of the study.With regard to slow transcranial magnetic stimulation aimed at resistant auditory hallucinations no significant adverse events have been disclosed. In a double blind study in which the left or right temporoparietal cortex was stimulated repeatedly for two weeks, subjects reported headache (N = 5), dizziness (N = 2), and amnesia (N = 1), while subjects in the sham arm of the study reported headache (N = 2), dizziness (N = 1), and difficulty in concentrating (N = 1). These adverse effects disappeared within 10 min of the completion of each rTMS treatment and were seen with both left and right hemisphere treatment.

In accordance with clinical studies, the rodent studies available so far support the notion that rTMS is a safe technique even when used chronically, i.e. up to 11 weeks in rats. The use of rTMS in humans is regarded as safe.

Regarding deep TMS, a study of 35 healthy volunteers conducted in collaboration of Shalvata Mental Health Care Center, Sheba Medical Center and Neurobiology Department of Weitzman Institute of Science, has demonstrated the safety of deep TMS treatment. The study is enclosed.

In this study Deep TMS will be administered by a trained doctor, and all patients will wear ear-plugs as to avoid hearing damage.

Rationale

The rational of this study is based on the following :

Resistance to treatment , significant subjective suffering & risk of suicide

1. As mentioned earlier auditory hallucinations are reported by 50%-70% of patients with schizophrenia, most of whom, indeed, are successfully treated with antipsychotic medication, but 25%-30% of whom are refractory to antipsychotic drugs.
2. Auditory hallucinations can cause great distress, functional disability, and lack of behavioral control.
3. A variety of psychosocial treatments have been used, but their efficacy has been described mainly in individual case reports and their relative merits are unclear.
4. Falloon and Talbot (1981) reported that more than quarter of their schizophrenic patients had made a serious suicide attempt in response to auditory hallucinations.

Promising response of auditory hallucinations to TMS

* A double blind study of Thirty-nine patients with schizophrenia with treatment-refractory auditory hallucinations showed that daily repetitive TMS at 1 Hz for 20 min per day for 10 treatment days over the left or right temporoparietal achieved significant changes in the frequency of auditory hallucinations, positive symptoms of PANSS, and CGI-I.
* Transcranial Magnetic Stimulation of Left Temporoparietal Cortex in frequency of 1 Hz for 9 days in 24 patients with schizophrenia /schizoaffective disorder and medication-resistant auditory hallucinations achieved substantial improvement in hallucinations frequency and attentional salience with 52% of patients maintaining improvement for at least 15 weeks.
* A study of 24 patients with schizophrenia given low frequency (1 Hz) repetitive transcranial magnetic Stimulation to the left temporoparietal cortex over 5 consecutive working days achieved improvement in Auditory Hallucinations Rating Scale scores as well as in source monitoring (= increased ability in identifying self-generate items as having come from themselves).
* A double-blind crossover study in ten schizophrenia patients with resistant auditory hallucinations given 5 days of low frequency rTMS (1 Hz) over the left temporoparietal cortex demonstrated a diminution of 56% of the hallucinations as reflected in reduction in all seven items of the auditory hallucinations rating scale as well as a diminution in SAPS scores.

Reasons to believe that right frontotemporal TMS stimulation cortex can ameliorate auditory hallucinations include evidence that right temporoparietal stimulation achieved significant changes in the frequency of auditory hallucinations,in the patients with auditory hallucinations an increase in blood flow is noted in the right superior temporal gyrus, right temporal lobe activation during auditory hallucination, effect of rTMS can spread to the opposite hemisphere through interhemispheric connections,some evidence that brain circuits involved in the production of auditory hallucinations and symptoms of schizophrenia are widespread and not confined in the left temporoparietal cortex.

Advantages of deep TMS over non-deep TMS

Deep TMS can reach brain structures as deep as 5 cm whereas non-deep TMS can reach structures less than half that distance. As deep brain structures such as thalamic, limbic and paralimbic regions have been shown to be activated during auditory hallucinations and suspected to play a role in the pathogenesis of auditory hallucinations, their stimulation may attenuate auditory hallucinations. Non-deep TMS can stimulate the cortex but not the neuronal pathways connecting it to deeper brain structures and which stimulation may be additive. According to Cleghorn et al the striatum plays a critical role in auditory hallucinations.

Methods

Each site is intended to recruit 20 patients aged 18-60 years old, diagnosed as suffering from schizophrenia and experiencing auditory hallucinations on daily basis. The operator as well as the rater will be blind to the kind of treatment being given to the specific patient they treat/evaluate clinically. Patients will be randomly and equally divided to 2 study groups:

Group 1:

10 patients will be given 20 minutes stimulation with real deep H1-Coil TMS to the Left Temporo-parietal Cortex in frequency of 1 Hz with 120% motor threshold during 20 consecutive working days.

Group 2:

10 patients will be given 20 minutes stimulation with sham deep H1-Coil TMS to the Left Temporo-parietal Cortex in frequency of 1 Hz with 120% motor threshold during 10 consecutive working days, and thereafter 20 sessions of real TMS with the same parameters (=Left Tempor-oparietal Cortex in frequency of 1 Hz with 120% motor threshold).

Schedule of Patient evaluation

Patients will be evaluated by the following manner:

Group 1:

Within 72 hours before first TMS study session , 24 hours after 10th session, right before the 11th session and again 24 hours after 20th session, one week after last session and one month after last session.

Group 2:

Within 72 hours before first TMS study session , 24 hours after 10th session, right before the 11th session and again 24 hours after 20th session right before the 21th session, 24 hours after 30th session ,one week after last session and one month after last session.

Patients' evaluation will include the following measures:

1. Auditory hallucinations Rating Scale developed by Hoffman and colleagues (2003).
2. Scale for the Assessment of Positive Symptoms scores (SAPS; Andreasen and Olsen 1982).
3. Clinical Global Impressions (CGI).
4. Assessment of Negative Symptoms (SANS).
5. Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q ).
6. Quick Inventory of Depressive Symptomatology ( QIDS-SR16 )
7. Personal and Social Functioning (GAF)
8. The magnitude of auditory hallucinations will be evaluated in every patient by his closest care taker according to the care taker impression of the patient's behavior (For example talking to himself), acts which the patient explains as being an obedience to the "voices'" commands or an attempt to lessen the voices (For example not leaving home due to fear of voices escalation), or being unresponsive to care takers questions or orders due to distraction by hallucinations. The care taker evaluation will take place one week prior to first TMS session, continuing on daily basis until one week after the last TMS session. This evaluation will hence be called "Care taker auditory hallucinations evaluation" or CTAHE. The care taker will evaluate the patient's hallucinatory behavior on a scale from 0 to 10, in which "0" is completely hallucination free and "10" being behavior dictated by hallucinations alone.This could be done using a visual analogue scale.

Average ratings can later be compared between pre & post treatment periods. As the care taker will be blind to TMS given to the patient (sham or real) and A care taker "Placebo" impression can be thus overcome. Clinical response will be judged according Hoffman's definition of positive response (50% or greater improvement in the auditory hallucinations scores)

Inclusion criteria

* Patients will fulfill DSM-IV-TR diagnostic criteria for schizophrenia
* Patients reporting auditory hallucinations on average at least 5 times per day based on prospective assessment using a diary or handheld counter.
* Patients are maintained on their psychotropic medication at steady dosages for at least 4 weeks before study entry and for the duration of the trial.

Exclusion criteria

Cardiac pacemaker implant, or a history of epilepsy, neurosurgery, or brain trauma patients suffering from chronic medical conditions of any sort, history of current hypertension, history of seizure or heat convulsion, history of epilepsy or seizure in first degree relatives, history of head injury, history of any metal in the head (outside the mouth), known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips, or any medical pumps, history of frequent or severe headaches, history of migraine, history of hearing loss, known history of cochlear implants, history of drug abuse or alcoholism, pregnancy or not using a reliable method of birth control (non-pregnancy will be proved by beta-HCG test),, systemic and metabolic disorders, inadequate communication skills or under custodial care.

Informed consent

After receiving a full explanation of the procedures, all subjects signed a written informed consent statement approved by the Helsinki Ethics Committee of Beer-Yacoob Mental Health Center.

Manual Explanation and information for Patient use

Every patient will be served with a simple explanation regarding the study aims and importance as well as possible risks and inconveniences as a result of magnetic stimulation.

Physical evaluation prior to and after study

In addition to the clinical follow up mentioned above, patients will undergo blood pressure, pulse rate, general physical examination (Beer-Yaacov physical examination on admission to hospitalization version), ECG prior to treatment as well as after the last session.

ELIGIBILITY:
Inclusion Criteria:

* Patients will fulfill DSM-IV-TR diagnostic criteria for schizophrenia
* Patients reporting auditory hallucinations on average at least 5 times per day based on prospective assessment using a diary or handheld counter.
* Patients are maintained on their psychotropic medication at steady dosages for at least 4 weeks before study entry and for the duration of the trial.

Exclusion Criteria:

* Cardiac pacemaker implant, or a history of epilepsy, neurosurgery, or brain trauma patients suffering from chronic medical conditions of any sort
* History of current hypertension
* History of seizure or heat convulsion
* History of epilepsy or seizure in first degree relatives
* History of head injury
* History of any metal in the head (outside the mouth)
* Known history of any metallic particles in the eye
* Implanted cardiac pacemaker or any intra-cardiac lines
* Implanted neuro-stimulators
* Surgical clips or any medical pumps
* History of frequent or severe headaches
* History of migraine
* History of hearing loss
* Known history of cochlear implants
* History of drug abuse or alcoholism
* Pregnancy or not using a reliable method of birth control (non-pregnancy will be proved by beta-HCG test)
* Systemic and metabolic disorders
* Inadequate communication skills or under custodial care.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
1.Auditory hallucinations Rating Scale developed by Hoffman and colleagues (2003) 2.SAPS 3.CGI 4.SANS 5.GAF | Prospective

SECONDARY OUTCOMES:
Q-LES-Q | prospective
  Quality of Life Enjoyment and Satisfaction Questionnaire
QIDS-SR16 | prospective
  Quick Inventory of Depressive Symptomatology
CTAHE | prospective
  The care taker evaluation will take place one week prior to first TMS session, continuing on daily basis until one week after the last TMS session. This evaluation will hence be called "Care taker auditory hallucinations evaluation" or CTAHE. The care taker will evaluate the patient's hallucinatory behavior on a scale from 0 to 10, in which "0" is completely hallucination free and "10" being behavior dictated by hallucinations alone.

CONTACTS AND LOCATIONS:
Overall Officials: Oded Rosenberg, M.D., Principal Investigator — Beer Yaakov Mental Health Center
Locations (1):
- Beer-Yaacov MHC, Beer Yaacov, Israel, Israel

REFERENCES:
- [Derived] Rosenberg O, Gersner R, Klein LD, Kotler M, Zangen A, Dannon P. Deep transcranial magnetic stimulation add-on for the treatment of auditory hallucinations: a double-blind study. Ann Gen Psychiatry. 2012 May 6;11:13. doi: 10.1186/1744-859X-11-13. PMID 22559192
- [Derived] Rosenberg O, Roth Y, Kotler M, Zangen A, Dannon P. Deep transcranial magnetic stimulation for the treatment of auditory hallucinations: a preliminary open-label study. Ann Gen Psychiatry. 2011 Feb 9;10(1):3. doi: 10.1186/1744-859X-10-3. PMID 21303566